CLINICAL TRIAL: NCT06505798
Title: Cryoballoon/Radiofrequency/Pulsed Field Ablation of Atrial Fibrillation Versus Medical Treatment for Heart
Acronym: CRAAFT-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 136905; CS/F/21/190034 CRAAFT-HF (Other Grant/Funding Number: British Heart Foundation); 281142 (Registry Identifier: IRAS project ID); 24/LO/0301 (Other: London - Hampstead Research Ethics Committee)
Record Dates: First submitted 2024-07-01; First posted 2024-07-17 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation (AF)
Keywords: AF
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: This is a randomised, adaptive open label multicentre clinical trial which compares optimal medical therapy (as per standard of care) with catheter ablation plus optimal medical therapy alone in participants with HfrEF (LVEF<50%) and paroxysmal or persistent atrial fibrillation.
  This design is adaptive in that the required sample size is reviewed in an interim analysis at 80% recruitment. This interim analysis aims to ensure that sufficient patients are recruited to maintain the conditional power of the study at 80% or higher. Options which can be deployed at the interim analysis include increasing patient numbers and increasing duration of follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The optimal medical therapy as per standard of care (No Intervention): Participants randomised to the optimal medical therapy arm will receive optimal medical therapy according to the most contemporary ESC HF guidelines.
- The catheter ablation (Other): Catheter ablation is an established therapeutic strategy in patients without HF that aims to convert AF to sinus rhythm in symptomatic, drug-refractory AF in patients.
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Catheter Ablation — Participants randomised to the catheter ablation arm will undergo Pulmonary Vein Isolation (PVI) which is the essential ablation intervention. The technique used will be at the discretion of the treating physician but may include Cryoballoon (Medtronic/Boston Scientific), Radiofrequency: CARTO (Biosense), pulsed field radiofrequency ablation, or Precision (Abbott Medical) electro-anatomical mapping systems. Additional ablation lesions may be delivered as preferred by the operator and will be documented. Electro-anatomical voltage maps will be collected (in SR/AF) and stored for later analysis.
  Arms: The catheter ablation

SUMMARY:
Atrial fibrillation (AF) is a common heart rhythm disorder that causes an irregular heart beat and is a cause of heart failure (HF). Treatments include drugs to slow the heart rate, anti-arrhythmic drugs or ablation of the heart to help preserve normal rhythm. A number of trials have suggested that ablation may be superior to drug treatment to reduce hospitalisations or prevent early death. However, these studies have been small and the results not applicable to the general population with AF and heart failure in the UK. This international study will compare catheter ablation and optimal medical therapy versus optimal medical therapy alone to see if catheter ablation reduces unplanned heart failure hospitalisations and death rates and improves quality of life.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) increases the severity of, and death from, heart failure (HF). Several small studies have demonstrated that restoration of sinus rhythm by catheter ablation in patients with HF improves left ventricular (LV) function and exercise tolerance. What is unknown is whether or not AF ablation reduces all-cause death and urgent CV hospitalisations in populations with HF. The current trial will answer this outstanding question, which is faced by HF clinicians and electrophysiologists on a daily basis. AF ablation can be performed very effectively and efficiently using a cryo-balloon or radio-frequency ablation PVI technique. These techniques have evolved slowly and are unlikely to change substantially over the course of this trial. One small trial (n=363) in implantable cardioverter-defibrillator and CRT defibrillator recipients (CASTLE-AF) reported a death benefit of AF ablation but the patients were highly selected and the death reduction was far higher than real world expected differences. Recent studies have noted that the population randomised in CASTLE-AF was not representative of the general HF population with only 7% of patients in the "real world" setting meeting the trial entry criteria. CASTLE-AF is therefore provocative but inconclusive; it has made little change to clinical practice. As no studies have investigated the death benefit in a general HF population, the proposed trial is necessary and warranted. This study is designed as a randomised, open label multicentre clinical trial in which catheter ablation and medical therapy is compared to medical therapy alone in patients with HF with reduced ejection fraction (<50%) and paroxysmal or persistent AF to determine if this reduces all-cause death and urgent CV hospitalisations as well as improving QoL. By utilising the clinical and research networks of the British Heart Failure Society and British Heart Rhythm Society (BHRS) we will recruit 1200 patients. The current trial will be almost three times the size of the only previous inconclusive trial which was reported in the New England Journal of Medicine.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged ≥18 years.
2. Patient is willing and able to give informed consent for participation.
3. Able and willing to comply with all study requirements, including ability to participate in study for 12 months.
4. Willing to allow their General Practitioner (GP) to be notified of participation in the study.
5. Patient with one of the following AF categories and at least one episode of AF documented (by any means eg ECG, Holter, Cardiac Implantable Electronic Device (CIED) interrogation or any other means):

   * Paroxysmal AF defined as spontaneous self-terminating AF lasted > 6 hours and <7 days.
   * Persistent AF as defined by at least one episode of AF >7 days but not >3 years (since 1st documentation)
6. Optimal tolerated medical therapy for HF (including ACE-I (or ARB or ARNi), beta-blocker, SGLT2 inhibitor and mineralocorticoid receptor antagonist (MRA) and cardiac resynchronisation therapy (CRT) where indicated & tolerated) for at least 6 weeks (according to the most contemporary European Society of Cardiology (ESC) HF guidelines). Maximal doses of these drugs are not mandated.
7. New York Heart Association Classification (NYHA) class II to III
8. LVEF <50% (Cardiac imaging report of LVEF<50% within 1 year (by echocardiography, cardiac magnetic resonance imaging or nuclear cardiology assessment)) AND after optimisation of medical therapy (see previous definition). Note - a LVEF of <50% must be documented by any cardiac imaging performed after optimisation of medical therapy. Documentation of other baseline echocardiographic parameters (eg LA volume, E/E' etc can be obtained from any echocardiogram within 2.5 years). This allows a handheld or echocardiogram focused on LVEF assessment.

   1. For those with LVEF 41-49% and without ongoing atrial fibrillation/flutter, N-terminal pro B-type natriuretic peptide (NT-proBNP) of ≥300pg/mL is required within 12 months prior to randomisation.
   2. For those with LVEF 41-49% and with ongoing atrial fibrillation/flutter, NTproBNP of ≥600pg/mL is required within 12 months prior randomisation.
   3. For those with LVEF ≤40%, NTproBNP is not required

Exclusion criteria:

1. Long standing (>3 year) persistent or permanent AF.
2. Previous atrioventricular (AV) nodal ablation.
3. Previous pulmonary vein isolation (PVI) or surgical ablation.
4. Recent (<90 days) (type 1 spontaneous) myocardial infarction (type 2 myocardial infarctions are not an exclusion criterion), percutaneous coronary intervention, coronary artery bypass grafting, cardiac resynchronisation therapy or stroke.
5. Severe aortic or pulmonary valve disease.
6. Severe primary or secondary mitral valve regurgitation.
7. Active illness (other than HF) likely to result in death within 2 years.
8. People who are pregnant or planning to become pregnant during the trial.
9. People who are breastfeeding.
10. Known allergy to contrast.
11. Contraindication for PVI.
12. Other conditions that may prevent subjects from adhering to the trial protocol, in the opinion of the investigator.
13. Currently participating in another randomised controlled trial of another drug or medical device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2031-12-15 (Estimated); Study Completion 2031-12-15 (Estimated)

PRIMARY OUTCOMES:
Time to first all-cause death and urgent CV hospitalisation | 2 years minimum (range: 2-5.5 years)
  The primary outcome (time to first all-cause death and urgent CV hospitalisation) will be summarised by randomised group and analysed using a Cox proportional hazards regression model for time to first event, adjusting for factors used to balance the randomisation.

SECONDARY OUTCOMES:
Total (first and recurrent) all-cause death and urgent cardiovascular hospitalisations. | 2 years minimum (range: 2-5.5 years)
  Total (first and recurrent) number of all-cause deaths and urgent cardiovascular-related hospitalisations. Joint frailty models will be used to analyse time to death and recurrent urgent CV hospitalisations simultaneously. Additionally, negative binomial regression will be used to analyse the number of recurrent urgent CV hospitalisations.
QoL at 6 and 12 months assessed using the KCCQ-CSS. | 12 months
  Quality of Life (QoL) at 6 and 12 months assessed using the Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS). Linear mixed effects regression models will be used to analyse repeated measurements of QoL. Scored from 0- 100, with a higher score indicating better health.
Time to all-cause death | 2 years minimum (range: 2-5.5 years)
  Time to all-cause death will be analysed using Cox proportional hazards regression model for time to event, matching the primary outcome.
Total (first and recurrent) all-cause death and urgent HF hospitalisations | 2 years minimum (range: 2-5.5 years)
  Total (first and recurrent) number of all-cause deaths and urgent heart failure-related hospitalisations. Joint frailty models will be used to analyse time to death and recurrent urgent HF hospitalisations simultaneously. Additionally, negative binomial regression will be used to analyse the number of recurrent urgent HF hospitalisations.
Cardiovascular death | 2 years minimum (range: 2-5.5 years)
  Total number of cardiovascular-related deaths. Cox proportional hazards regression model for time to event, matching the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pier Lambiase, Principal Investigator — University College, London; Mark Petrie, Principal Investigator — University of Glasgow
Locations (14):
- United Kingdom (14):
  - Mid and South Essex NHS Foundation Trust, Basildon
  - University Hospitals Dorset NHS Foundation Trust, Bournemouth
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Golden Jubilee National Hospital, Glasgow
  - Hull University Teaching Hospitals NHS Trust, Hull
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Royal Brompton and Harefields Hospitals, London
  - Barts Health NHS Trust, London
  - Imperial College Healthcare NHS Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Nottingham University Hospital NHS Trust, Nottingham
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Swansea Bay University Health Board, Swansea